CLINICAL TRIAL: NCT02861196
Title: Research on the Combined-Modality Treatment Model of Bladder Preservation in Muscular Invasive Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianzhong Shou, Clinical Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC 2015L12
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Cystectomy

ARMS (1):
- Therapy Arm (Experimental): Patients who have response to neoadjuvant chemotherapy will be separated into two groups (GI cT0-1 and G2 ≥cT2). G1receive concurrent radiochemotherapy, and G2 receive partial resection of the bladder+lymphadenectomy+adjuvant radiotherapy.Patients who have no response to neoadjuvant chemotherapy or disagree to receive the sequential treatment will receive the radical resection of bladder.
  Interventions: Procedure: Intensity modulated radiation therapy, Radical cystectomy

INTERVENTIONS:
Procedure: Intensity modulated radiation therapy, Radical cystectomy — Postoperative Intensity modulated radiation therapy(IMRT) will be applied to effective team.Radical cystectomy will be applied to ineffective team.

SUMMARY:
This research aims to explore the therapeutic effect of neoadjuvant chemotherapy in muscular invasive bladder cancer of T2-4aN0M0, and the survival effect of combined-modality treatment model，then to clarify the probability of bladder preservation, corresponding cancer specific survival, and the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. bladder urothelium carcinoma
2. cT2-4aN0M0
3. life expectancy≥1 year
4. ECOG PS 0-1
5. have no previously received radiotherapy or chemotherapy
6. have no major organ dysfunction
7. have been provided informed written consent

Exclusion Criteria:

1. extensive carcinoma in situ or ureter invaded
2. distant metastasis at primary diagnosis or lymphatic metastasis according to clinical diagnosis
3. have severe major organ dysfunction
4. cannot finish treatments because of other severe diseases or life expectance≤6 months
5. exist other malignant tumors
6. have severe coagulation disorders
7. no other trails participated in 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
bladder preservation rate | 3 years
  bladder preservation rate

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Shou, MD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China